CLINICAL TRIAL: NCT01834950
Title: Identification of Early Markers of Response and Resistance to Trastuzumab in Patients With Localized Human Epidermal Growth Factor Receptor-2(HER-2)-Positive Breast Cancer Candidates for Breast Conserving Surgery
Brief Title: Identification of Early Markers of Response and Resistance to Trastuzumab
Acronym: HERBIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012-A01364-39; 2012/1909 (Other: CSET number)
Record Dates: First submitted 2013-03-01; First posted 2013-04-18 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Untreated Human Epidermal Growth Factor Receptor-2(HER2)Positive Early Breast Cancer
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trastuzumab (Experimental): The study is a single arm prospective study, aiming at identifying biomarkers of early response to trastuzumab
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test

SUMMARY:
The study is a single arm prospective study, aiming at identifying biomarkers of early response to trastuzumab. It is a prognostic factor study recruiting all consecutive cases of HER-2 positive breast cancer eligible for a pre-operative treatment by trastuzumab, followed by breast conserving surgery. The investigators will study the association between the value of biomarkers measured at diagnosis and the Response Evaluation Criteria in Solid Tumors response (partial and complete response) using a logistic regression (main analysis).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Female patients aged 18 years or older.
* Histologically or confirmed untreated invasive carcinoma of the breast
* Previous treated invasive breast carcinoma or ductal carcinoma in situ are allowed, assuming there is no evidence of disease at the moment of the inclusion in the protocol, and patients are not on any current treatment
* Candidates for breast conserving surgery: patients with a minimum size of 11 mm measured by breast US. Bilateral and multifocal tumors are allowed, assuming the biopsies pre- and post-treatment are performed in the same target lesion.
* HER2-positive (defined as either immunohistochemistry [immuno-histochemistry ] 3+ or in situ hybridization [ISH] positive) as assessed by local laboratory on primary tumor (ISH positivity is defined as a ratio of 2.2 or greater for the number of HER2 gene copies to the number of signals for abnormality on chromosome 17 (CEP17), or for single probe tests, a HER2 gene count greater than 4) and/or by PCR.
* No evidence of metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0/1.
* Left ventricular ejection fraction (LVEF) of at least 50%
* Negative pregnancy test in women of childbearing potential (premenopausal or less than 12 months of amenorrhea post-menopause, and who have not undergone surgical sterilization).
* For women of childbearing potential who are sexually active, agreement to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception during and for at least 6 months post-treatment.
* Maximum time allowed between collect of the informed consent and first administration of treatment :21 days
* All patients candidates for initial surgery and not candidates for primary chemotherapy (T3 acceptable if multifocal and decision primary surgery).

Exclusion Criteria:

* Patients non-candidate for initial breast surgery or patient's candidate for neoadjuvant chemotherapy ;
* Patients receiving another concomitant anticancer treatment like chemotherapy, immunotherapy, anti-HER2 treatment other than trastuzumab, endocrine treatment, or radiotherapy ;
* Known hypersensibility to trastuzumab ;
* Serious uncontrolled concomitant disease that would contraindicate the use of trastuzumab or that would put the patient at high risk for treatment-related complications ;
* Inadequate organ function, evidenced by the following laboratory results:

  * Absolute neutrophil count <1,500 cells/mm3
  * Platelet count <100,000 cells/mm3
  * Hemoglobin <9 g/dL
  * Total bilirubin greater than the upper limit of normal (ULN) (unless the patient has documented Gilbert's syndrome)
  * Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) >2.5 x ULN
  * Serum creatinine >2.0 mg/dL or 177 μmol/L
  * International normalized ratio (INR) and activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) >1.5 x ULN (unless on therapeutic coagulation)
* Uncontrolled hypertension (systolic >150 mmHg and/or diastolic > 100 mmHg) or clinically significant (i.e. active) cardiovascular disease: cerebrovascular accident/stroke or myocardial infarction within 6 months prior to first study medication; unstable angina; CHF of New York Heart Association (NYHA) Grade II or higher; or serious cardiac arrhythmia requiring medication ;
* Current known infection with human immunodeficiency virus (HIV), hepatitis B or C virus ;
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol ;
* Pregnant or breastfeeding patients ;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-03-27 (Actual); Primary Completion 2017-12-10 (Actual); Study Completion 2017-12-10 (Actual)

PRIMARY OUTCOMES:
Response rate | assessed after 6 weeks
  The response after 2 cycles of 3-weekly trastuzumab will be assessed as per Response Evaluation Criteria in Solid Tumors(RECIST) 1.1 criteria and will be correlated with biomarkers.

SECONDARY OUTCOMES:
Pathological complete response | assessed after 6 weeks
  According to Chevallier's classification

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Gustave Roussy, Villejuif, Val De Marne, France